CLINICAL TRIAL: NCT00341458
Title: Breast, Ovarian and Endometrial Cancer Case-Control Study in Poland
Brief Title: Breast Cancer in Poland: An Expanded Study to Assess Occupational and Environmental Factors and Interactions With Genetics
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999040; OH99-C-N040
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms; Gonadal Disorders; Uterine Diseases
Keywords: Breast Cancer; Environment; Genetics; Epidemiology
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms; Gonadal Disorders; Uterine Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cancer Cases: Women 20-74 years old, residents of Warsaw and Lodz that were newly diagnosed with confirmed in situ or invasive breast cancer or ovarian or endometrial cancer

SUMMARY:
The Polish breast, ovarian and endometrial cancer study is a complex molecular epidemiologic study that is expected to enroll about 2,500 breast cancer, 450 ovarian and 450 endometrial cancer cases and 2,500 controls from Warsaw and Lodz, two major cities in Poland. This large population-based study combines state-of-the-art techniques of exposure assessment and collection of biological specimens to allow for the study of a wide range of biomarkers. Exposure information is obtained through detailed personal interviews, anthropometric measurements, physical activity monitors, and collection of dust samples from the participants homes. The collection of biological specimens includes blood samples processed as cryopreserved whole blood, serum+ blood clot, plasma+buffy coat+red blood cells; 12-hour overnight urine; paraffin embedded tumor and normal tissue; and fresh tissue from tumors, non-neoplastic breast tissue and mammary fat tissue. Subject enrollment started in June 2000 and is expected to continue until January 2003 for breast cancer cases and controls and June 2003 for ovarian and endometrial cancer cases. As of May 2002, we have identified 2,207 breast, 138 ovarian and 235 endometrial cancer cases and 2,327 controls. The response rates to the interview are 81% for breast, 90% for ovarian and 83% for endometrial cancer cases and 70% for controls. Most women who agree to the interview agree to provide biological specimens (about 90% of cancer cases and controls agree to provide a blood sample), anthropometric measurements (95% of breast cancer cases and controls) and wear a physical activity monitor (79% breast cancer cases and 90% of controls)....

DETAILED DESCRIPTION:
The Polish breast, ovarian and endometrial cancer study is a complex molecular epidemiologic study conducted in two major cities in Poland (Warsaw and Lodz) that enrolled 2,386 breast cancer cases and 2,503 controls, and is expected to enroll about 400 ovarian, 600 endometrial cancer cases and 600 additional controls by September 2004. This large population-based study combines state-of-the art techniques of exposure assessment and collection of biological specimens to allow for the study of a wide range of biomarkers. Exposure information is obtained through detailed personal interviews, anthropometric measurements, physical activity monitors, and collection of dust samples from the participants' homes. The collection of biological specimens includes blood samples processed as cryopreserved whole blood, serum+ blood clot, plasma+buffy coat+red blood cells; 12-hour overnight urine; paraffin embedded tumor and normal tissue; and fresh tissue from tumors, non-neoplastic breast tissue and mammary fat tissue. Subject enrollment started in June 1, 2000.The last day of diagnosis for eligible breast cancer cases was December 31, 2003. The final response rates to the interview for the breast cancer component of the study are 79% for breast cancer cases and 69% for controls. Among women who agree to the interview, most of them agree to provide biological specimens (84% of breast cancer cases and 92% of controls agree to provide a blood sample; 82% of cases and 89% of controls agree to provide a urine sample), anthropometric measurements (95% of breast cancer cases and 93% controls) and wear a physical activity monitor (76% of breast cancer cases and 84% of controls from the Warsaw study site). The final participation rates to the interview for the ovarian and endometrial component of the study are 78% for ovarian, 80% for endometrial cancer cases. Of these women, 85% of ovarian and 86% of endometrial cancer cases agreed to provide a blood sample. Urine samples, anthropmetric measurements, physical activity monitor data are not collected from ovarian and endometrial cases. We are currently working on the first manuscripts from the breast cancer component of the study. We have completed DNA extractions and the first genotype assays. In addition, we constructed tissue microarrays using formalin fixed tumor samples from breast cancer cases with invasive cancer and performed a number of immunohistochemical/immunofluorescence stains to evaluate etiologic heterogeneity of breast cancer risk factors by tumor type. For the ovarian/endometrial component of the study, we have completed the DNA extractions for all subjects, and incited the first analyses for endometrial study. Determination of the first genotypes for the ovarian/endometrial components and construction of tissue microarrays for endometrial cases is planned for 2005- 06.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cases for study will consist of all women ages 20-74 years who are newly diagnosed with either histologically or cytologically confirmed in situ or invasive breast cancers during the two and a half year study period.

In both Warsaw and Lodz, controls will be selected using the Polish Electronic System of Population Evidence localized in Warsaw (PESEL).

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible cases were women 20-74 years old, residents of Warsaw and Lodz that were newly diagnosed with confirmed in situ or invasive breast cancer between Jan 2000-Jan 2003, or ovarian or endometrial cancer diagnosed between June 2001-Dec 2003. A Rapid Identification System (RIS) was used at participating hospitals to identify eligible cases, and a Cancer Registry in Warsaw was used to identify cases missed by the RIS. Population control subjects were selected using the Polish @@@Electronic System, a database with demographic information from all residents of Poland. A random sample of women was chosen to represent the age distribution of women who develop breast, ovarian or endometrial cancer during the study period. Control selection was done on a quarterly basis from Jan 2000-June 2004.@@@Controls identified through Sept 2003 were matched to breast cancer cases by city and age in 5-year categories. Endometrial and ovarian controls were identified from June 2001-June 2004.
Sampling Method: Probability Sample
Enrollment: 6086 (Actual)
Dates: Start 1999-09-01 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Breast cancer | incident
  Pathologically confirmed diagnosis of breast cancer
Ovarian cancer | incident
  Pathologically confirmed diagnosis of ovarian cancer
Endometrial cancer | incident
  Pathologically confirmed diagnosis of endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Garcia-Closas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- Poland (2):
  - Nofer Institute of Occupational Medicine, Lodz
  - Maria Sklodowska Curie Memorial Cancer Center and Institute of Oncology, Warsaw

REFERENCES:
- [Background] Garcia-Closas M, Brinton LA, Lissowska J, Chatterjee N, Peplonska B, Anderson WF, Szeszenia-Dabrowska N, Bardin-Mikolajczak A, Zatonski W, Blair A, Kalaylioglu Z, Rymkiewicz G, Mazepa-Sikora D, Kordek R, Lukaszek S, Sherman ME. Established breast cancer risk factors by clinically important tumour characteristics. Br J Cancer. 2006 Jul 3;95(1):123-9. doi: 10.1038/sj.bjc.6603207. Epub 2006 Jun 6. PMID 16755295
- [Background] Garcia-Closas M, Brinton LA, Lissowska J, Richesson D, Sherman ME, Szeszenia-Dabrowska N, Peplonska B, Welch R, Yeager M, Zatonski W, Chanock SJ. Ovarian cancer risk and common variation in the sex hormone-binding globulin gene: a population-based case-control study. BMC Cancer. 2007 Apr 5;7:60. doi: 10.1186/1471-2407-7-60. PMID 17411440
- [Background] Garcia-Closas M, Egan KM, Newcomb PA, Brinton LA, Titus-Ernstoff L, Chanock S, Welch R, Lissowska J, Peplonska B, Szeszenia-Dabrowska N, Zatonski W, Bardin-Mikolajczak A, Struewing JP. Polymorphisms in DNA double-strand break repair genes and risk of breast cancer: two population-based studies in USA and Poland, and meta-analyses. Hum Genet. 2006 May;119(4):376-88. doi: 10.1007/s00439-006-0135-z. Epub 2006 Feb 17. PMID 16485136
- [Background] Brinton LA, Sakoda LC, Lissowska J, Sherman ME, Chatterjee N, Peplonska B, Szeszenia-Dabrowska N, Zatonski W, Garcia-Closas M. Reproductive risk factors for endometrial cancer among Polish women. Br J Cancer. 2007 May 7;96(9):1450-6. doi: 10.1038/sj.bjc.6603731. Epub 2007 Apr 10. PMID 17426703